CLINICAL TRIAL: NCT05013567
Title: Randomized, Double-Blind, Parallel, Phase III Superiority Clinical Trial to Evaluate the Efficacy and Safety of Ibuprofen Gel Compared With Placebo in the Treatment of Acute Musculoskeletal Pain
Brief Title: Efficacy and Safety Study of Ibuprofen Gel Compared to Placebo in the Treatment of Acute Musculoskeletal Pain
Acronym: PROGEL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brainfarma Industria Química e Farmacêutica S/A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HYP 001-21
Record Dates: First submitted 2021-08-03; First posted 2021-08-19 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2021-08

CONDITIONS: Musculoskeletal Pain; Acute Pain; Stretch; Sprains
Keywords: ibuprofen; ibuprofen gel; pain
MeSH Terms: conditions — Musculoskeletal Pain; Acute Pain; Sprains and Strains; Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen gel 5% (Experimental)
  Interventions: Drug: Ibuprofen gel
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ibuprofen gel — Ibuprofen gel 5% topically four times a day
  Arms: Ibuprofen gel 5%
Other: Placebo — Placebo gel topically four times a day
  Arms: Placebo

SUMMARY:
Phase III clinical trial, multicentre of superiority, randomized, double-blind, parallel groups, placebo-controlled and use of ibuprofen gel in the treatment of acute pain.

DETAILED DESCRIPTION:
This study is designed for the relief of acute musculoskeletal pain, characterized by pain in muscles, ligaments, tendons, and nerves.

It is performed in participants of both sexes, over 18 years of age, who have pain of moderate intensity as a result of ankle sprains, upper limb contusions, thigh muscle strains, or torticollis.

The rationale for studying the topical use of ibuprofen is the possibility of an alternative treatment for musculoskeletal pain, avoiding systemic adverse events caused by oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Have signed the informed consent form;
* Participants of both genders aged ≥ 18 years;
* Present acute musculoskeletal pain as a result of: ankle sprains, upper limb contusions, thigh muscle sprains, or torticollis;
* Present pain of moderate intensity by VAS scale (3 ≤ VAS ≤ 7);
* Pain onset time is less than 36 hours;
* Present intact skin at the trauma site;
* Participants of both sexes with the potential to become pregnant must be truly abstinent or use a highly effective method of contraception throughout the period of 30 days before the administration of the drug until 30 days after the end of treatment;
* Agree to safety laboratory tests: pregnancy test, complete blood count, and biochemical profile;
* Be able to understand the nature and purpose of the trial, including the risks and adverse events.

Exclusion Criteria:

* Participants under the age of 18;
* Participants with musculoskeletal pain as a result of fractures or dislocations;
* Participants with mild pain (VAS < 3) at the time of selection;
* Participants with severe pain (VAS > 7) at the time of selection;
* Participants with pain onset time greater than 36 hours;
* Participants with a history of chronic pain and acute pain spikes;
* Participants with loss of skin integrity at the trauma site;
* Have a known hypersensitivity reaction to the trial medication or chemically related compounds;
* Have a prior history of the following comorbidities: asthma or other allergic conditions, uncontrolled heart failure, chronic kidney disease, chronic liver disease, active peptic ulcer disease, or gastrointestinal bleeding;
* Suspect for COVID-19 according to the criteria defined by the World Health Organization;
* Regular use of analgesics, non-steroidal analgesics or anticoagulants;
* Use of oral or topical corticoids in the injured area;
* Being on medications that have relevant interactions with the trial drugs, such as non-steroidal anti-inflammatory drugs (NSAIDs), warfarin, lithium, methotrexate, acetylsalicylic acid, corticosteroids, oral hypoglycemic agents, beta blockers, angiotensin-converting enzyme inhibitors, antihypertensive agents, and diuretics such as furosemide or thiazide;
* Have had oral or topical analgesic treatment, including use of non-steroidal analgesics, within 72 hours prior to the screening visit;
* Participants using traditional Chinese or Japanese therapy (acupuncture);
* Abusive use of alcoholic beverages;
* Women who are pregnant, breastfeeding, planning to become pregnant, or who test positive for pregnancy during the trial period;
* Have participated in a clinical trial within the last 12 months;
* Have any condition that would preclude participation in the trial in the physician's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Superiority of ibuprofen gel over placebo in the treatment of acute musculoskeletal pain. | 5 days of treatment
  The primary endpoint of the study is the proportion of participants achieving at least 50% pain reduction on day 5 of treatment by assessing pain intensity using the Visual Analog Scale (VAS), compared to baseline VAS. (Scale = 0 to 10; 0 = mild pain and 10 = severe pain)

SECONDARY OUTCOMES:
Pain relief with study medication on days 3, 5, and 7. | 3, 5 and 7 days of treatment
  Pain relief by the adapted Pain Relief (PAR) Scale, with the 5 categories: 0 - no relief, 1- slight relief, 2 - moderate relief, 3 - considerable relief, and 4 - complete relief, on days 3, 5, and 7.
Interference of pain on physical activity on days 3, 5 and 7 | 3, 5 and 7 days of treatment
  Pain interference with physical activity by 4-point scale: 0 - no interference with physical activity; 1 - no restriction of physical activity, although some pain on movement; 2 - some restriction of physical activity, but not enough to prevent normal activity; 3 - unable to perform normal activities and with substantial limiting effects, on days 3, 5, and 7.
Time needed for pain improvement. | Through study completion, an average of 7 days
  Time needed for pain improvement (reduction of at least 50% of pain on the VAS scale)
Obtain the overall assessment of effectiveness, performed by the participant at the end of the treatment. | Through study completion, an average of 7 days
  Overall assessment of treatment by participant using 5-point scale: bad, fair, good, very good, and excellent.
Obtain the overall efficacy evaluation, performed by the investigator at the end of the treatment. | Through study completion, an average of 7 days
  Overall assessment of treatment by physician using 5-point scale: bad, fair, good, very good, and excellent.
Number of participants using rescue medication. | Through study completion, an average of 7 days
Time to use of rescue medication. | Through study completion, an average of 7 days

OTHER OUTCOMES:
Occurrence of adverse events (AEs) during the study period. | Through study completion, an average of 7 days
  Rate of occurrence of serious and non-serious AEs, related and unrelated to treatment groups throughout the clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Brainfarma Indústria Química Farmacêutica, Study Director — Brainfarma Industria Química e Farmacêutica S/A